CLINICAL TRIAL: NCT04888182
Title: The Effect of High Protein Diet in Combination With Physical Activity in the Rehabilitation of Patients With Chronic Obstructive Pulmonary Disease (COPD) at Risk of Malnutrition- a Pilot Study
Brief Title: High Protein Diet and Physical Activity in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, Primary Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBH-KU 33
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized, parellel, not blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): Individual nutritional guidance of a protein intake of ≥25 E%.
  Interventions: Dietary Supplement: intervention
- control (No Intervention): Free diet

INTERVENTIONS:
Dietary Supplement: intervention — a protein intake of ≥25 E%. An oral nutritional supplement (containing 1570 kJ/100 g and 92 g protein/100 g. Atpro 200) was used as supplement to the patients' habitual diet.
  Arms: intervention

SUMMARY:
COPD outpatients with severe and very severe (grade III-IV) disease at risk of malnutrition commencing rehabilitation (7-10-week physical activity program) were randomized to receive a high protein diet (≥ 25 energy percentage) or standard care.

DETAILED DESCRIPTION:
Peripheral muscle function was measured by 6MWD (6-meter-walk-distance) and handgrip strength; FFM was measured by bioimpedance, mid upper arm circumference, and mid-thigh circumference; quality of life was measured by CAT (????); and dyspnoea was measured by the Medical Research Council dyspnoea scale and Borg scores at baseline and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed COPD stage III or stage IV
* Nutritional risk by screening (NRS-2002)(Kondrup et al, 2002) and/or low-fat free mass (FFMI) (≤ 15% for women and ≤ 16% for men) measured by Bioelectrical Impedance Analysis (BIA)

Exclusion Criteria:

* Terminal phase of COPD
* Lung transplanted patients
* Severe Comorbidities influenzing the end-points (pancreatic insufficiency, severe hepatic failure, inflammatory gastrointestinal disease)

  * Multiple sclerosis
  * Any unwillingness or inability (e.g. not able to make notes of their nutritional intake, come to consultations or manage oral intake)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6MWD) | 7 weeks
  metres
hand grip strenght | 7 weeks
  kg

SECONDARY OUTCOMES:
Fat Free Mass (FFM) | 7 weeks
  Bioimpedance - kg
Dyspnoea after 6 minutes walk | 7 weks
  Medical Research Council (MRC) dyspnoea scale (scores range from 0 to 5)
Quality of life | 7 weeks
  self-administered COPD Assessment Test (CAT), 40-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Pulmonary Medicine, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mogelberg N, Tobberup R, Moller G, Godtfredsen NS, Norgaard A, Andersen JR. High-protein diet during pulmonary rehabilitation in patients with chronic obstructive pulmonary disease. Dan Med J. 2022 Oct 11;69(11):A03220185. PMID 36331152